CLINICAL TRIAL: NCT02914808
Title: Assessment of Tissue and Biomolecular Complements of Lower Limb Chronic Oedema
Brief Title: Oedema Study : Chroedem
Acronym: CHROEDEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL15_0489
Record Dates: First submitted 2016-09-02; First posted 2016-09-26 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lower Limb Chronic Oedema
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patients will undergo a lower limb MRI and blood tests

SUMMARY:
The chroedem study is aiming to assess tissue and biomolecular components of chronic lower limb oedema (CO). The investigators working hypothesis is that according to the aetiology of CO, the proportion of oedema & composition of peri-oedema tissues (fat, muscle, fibrosis/inflammation) might differ and could at least in part explain differences in failure/success of compressive therapies from one patient to another. For that purpose, 24 patients with a post-thrombotic syndrome (PTS)-related oedema and 24 patients with a primary lymphedema will undergo a magnetic resonance imaging (MRI)) of the legs and biological (genetic) testing.

DETAILED DESCRIPTION:
Chronic lower limb oedema is the consequence of an abnormal accumulation of fluid in the interstitium located beneath the skin of legs. It is a frequent disease with a significant morbidity (skin infections, leg ulcers…), which can deeply alter patient's quality of life.

On a pathological point of view, current main hypothesis is hemodynamic (i.e. failure of venous and lymphatic return).

Recent data suggest that other factors, particularly genetic ones (genes coding for proteins of inflammation or of fibrosis, for adipogenesis and for lymphangiogenesis…) could influence the development of CO. Stimulation of these mediators varies from one person to another and from one clinical setting to another (i.e. venous insufficiency vs. lymphedema etc…). One can therefore assume that CO is not a homogeneous entity and that the distribution of tissue components varies.

On a therapeutic point of view, this difference in the distribution of tissue components could at least in part explain the differences in effectiveness of compression therapy and in tissue dysmorphia from one person to another and from one type of CO to another.

The study primary objective is to assess and compare by MRI the different tissue components (oedema, fat, muscle, inflammation/fibrosis) of lower limb CO of venous vs. lymphatic origins.

The investigators shall conduct a prospective observational pilot study. 24 patients with a CO of PTS origin and 24 patients with a CO of lymphatic origin (primary lymphoedema) will undergo a clinical examination, 3-D laser scanner volumetry of their lower limbs, blood tests and a MRI of lower limb. Main exclusion criteria will be obesity and bilateral CO. The main primary outcome measure will be the proportion of fat, muscle and oedema assessed by MRI in a pre-determined lower limb area. The main secondary outcome measure will be the prevalence in each group of i) variations in exonic sequence of genes coding for proteins of inflammation/fibrosis, angiogenesis, adipogenesis; ii) variations in exonic sequence of genes reported in the literature as associated with primary lymphoedema.

This study should allow to better characterize tissue structure and inflammatory, adipous and angio-genetic profiles of lower limb CO. The potential therapeutic perspective is to adapt compressive therapies to the type of oedema and to test the impact of new therapies (e.g. anti-inflammatory drugs for oedema with important fibrotic component?).

ELIGIBILITY:
Inclusion criteria:

* Lower limb CO secondary to PTS or Primary lymphoedema (We will include secondary lymphedema of the lower limbs only if the matcing constraints on age and length of evolution do not allow pairing)

Exclusion criteria:

* Bilateral CO
* Obesity
* Mixed CO (PTS and lymphatic origins)
* CO of other origin : Heart failure, hepatic or renal impairment
* Denutrition
* Contra-indication to MRI
* Patient not affiliated to French Health Insurance System
* Patient protected by the law
* Patient refusing to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 patients with a CO of PTS origin and 24 patients with a CO of lymphatic origin (primary lymphoedema) will undergo a clinical examination, 3-D laser scanner volumetry of their lower limbs, blood tests and a MRI of lower limb. Main exclusion criteria will be obesity and bilateral CO.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of fat muscle and oedema assessed by MRI in a pre determined lower limb area | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: ISABELLE QUERE, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Pr Sophie BLAISE, Grenoble, Isère
  - University Hospital of Montpellier, Montpellier
  - University Hospital Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No